CLINICAL TRIAL: NCT04515355
Title: Preventing Job Loss Using Acceptance and Commitment Therapy in Vocational Rehabilitation
Acronym: MS-Proactive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NE20/130005
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with MS (PwMS) (Experimental): People with MS recruited to take part and will be randomised to receive the intervention of online programme of support.
  Interventions: Behavioral: Ready for MS
- People with MS (PwMS) - standard care (No Intervention): People with MS recruited to take part and will be randomised to receive the usual standard of care.

INTERVENTIONS:
Behavioral: Ready for MS — Receive 'ready for MS' programme in addition to standard care.
  Arms: People with MS (PwMS)

SUMMARY:
About 60-70% of people with multiple sclerosis (PwMS) lose employment within 10 years of the diagnosis. This can be due to complex personal and work-based factors including psychological factors. MS-PROACTIVE aims to test an online self-help therapy to support PwMS to stay in work called 'READY for MS'. This is a type of Acceptance and Commitment therapy. It is a way to provide treatment in a flexible way without people having to go to see a psychologist.

The aim of the treatment is to improve self-efficacy which has been shown to be a significant factor for helping PwMS who want to work to stay in work.

The research team will initially develop an online version of READY for MS. We will ask 4 PwMS to test the online'READY for MS' and provide feedback and advice on any necessary changes. We will then recruit and randomise 88 PwMS in Leeds and London who are at risk of job loss. Participants in the active treatment group will use the online treatment in addition to their usual care; the control group will receive their usual care. The participants will complete questionnaires at the start of the study, at 8 weeks and 6 months measuring time off work and work instability (to measure risk of job loss), self-efficacy, mood, quality of life, fatigue and the impact of MS. The questionnaire data will be analysed to test the effectiveness of the treatment. The research team will also interview 4 PwMS at each site at the start of the study, at 8 weeks and 6 months to find out about their experience of using READY for MS in more detail. This will help to inform the use of READY for MS in a larger trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Employed people with a confirmed diagnosis of multiple sclerosis. Paid employment including full-time or part-time work and self-employed. Age 18 years and over Access to a computer or tablet for the on-line sessions. Ability to complete questionnaires at three time points.

Exclusion Criteria:

* Unpaid employment eg voluntary work. PwMS who are planning to retire or fully leave employment in the time period of the RCT. On sick leave or maternity leave at the time of recruitment.

Significant cognitive impairment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Completing the Ready for MS programme | 7 weeks
  Ready for MS is an online programme of support and participants will comple 7 thirty minute online support sessions over 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom